CLINICAL TRIAL: NCT07016295
Title: Developing an Accessible, Cost-Effective Motion Analysis Tool for Arm Movement After Stroke
Brief Title: Monitoring Arm Recovery After Stroke (MARS)
Acronym: MARS
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LRS/RGO-24/25-47508
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: biomechanics; pose estimation models; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke survivors
  Interventions: Behavioral: Biomechanical analysis of arm movement; Behavioral: Pose estimation of arm movement
- Healthy age-matched controls
  Interventions: Behavioral: Biomechanical analysis of arm movement; Behavioral: Pose estimation of arm movement

INTERVENTIONS:
Behavioral: Biomechanical analysis of arm movement — Marker based kinematic analysis
Behavioral: Pose estimation of arm movement — Marker free kinematic analysis

SUMMARY:
People who have a stroke often find it hard to do the things they did before. This can be caused by problems with arm movement. One in five people do not get any arm movement back after a stroke.

Arm movements can be measured accurately in a laboratory, but it is very expensive and not easy to do in hospital. That means it is hard to tell if the arm is recovering to move like it did before the stroke or adapting to perform tasks in other ways.

To tell if a treatment is working, the investigators are making a phone app to record arm movement, using the camera. The recordings will be turned into data showing movement difficulties and sent to hospital records for clinicians. Clinicians will see if movement changes, to help choose the best treatment.

The investigators are looking for twelve stroke survivors to help test this app.

* The session will be at King's College London, on Guy's Campus.
* It will run for 2-3 hours.
* Participants will wear a vest or tight-fitting clothes.
* The investigators will place non-invasive markers on the participants arm.
* The investigators will video simple movements such as drinking from a cup.
* The investigators will also measure the same simple movements using the laboratory cameras.

This will show us if our app can measure arm movement as well as laboratory tests. If they do, the investigators will know the app is accurate.

In future this technology can improve recovery by correcting stroke survivors when they perform home exercises.

DETAILED DESCRIPTION:
Upper limb recovery after stroke remains poor and 20% of stroke survivors do not recover arm movement. To improve outcome and advance insights to recovery mechanisms, an international collaboration has proposed a standardised set of outcome measures, including movement kinematics. Kinematics are moresensitive to change than clinical measures and can differentiate whether recovery is achieved by compensating to impairment or true recovery. However, kinematic assessments are not performed in clinical practice as 3-D motion capture requires expensive equipment and expertise for set-up and analysis.

The investigators therefore aim to develop a low-cost tool to measure kinematics. Open-source Artificial Intelligence models can detect positions and orientations on video and are called pose estimation models. The objectives will be to deploy and test these models in stroke survivors. The investigators will invite 12 stroke survivors with mild to moderate upper limb impairment and compare the accuracy of the models to gold-standard kinematic analysis when performing a variety of upper limb tasks. The investigators will optimise the models in case of any discrepancies. The investigators will develop a front-end smartphone app to instruct, record and provide feedback of arm movement performance to clinicians and stroke survivors. The investigators will develop the software back-end performing analysis of recorded movements and integrating these findings into electronic healthcare records for longitudinal performance tracking.

This accessible technology will provide clinicians kinematic analyses. Kinematics can guide treatment modifications and progression to improve upper limb movement.

ELIGIBILITY:
Stroke survivors

Inclusion Criteria:

* History of stroke
* Arm impairment evidenced by Fugl-Meyer Upper Limb Assessment between 9-60/66.

Exclusion Criteria:

* Severe cognitive impairment preventing ability to consent to treatment and understand and follow research protocol
* Severe language deficit preventing ability to consent to treatment and understand and follow research protocol
* Shoulder pain >3/10 on visual analog scale
* Unable to maintain independent sitting balance without a high back support.
* Wheelchair users that are unable to transfer with assistance of 1 to lab chair or whose wheelchair backrest cannot colapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 stroke survivors 8 Healthy age-matched controls
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pose estimation model accuracy | During intervention
  Agreement between pose estimation and biomechanics measurements

SECONDARY OUTCOMES:
Fugl-Meyer Upper limb Assessment | baseline, before intervention
Motricity Index | baseline, before intervention
  Strength
Cancellation OCS | baseline, before intervention
  neglect
Box and block | during the intervention
  dexterity
ARAT-2 | during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vasa Curcin, PhD, Study Chair — King's College London
Locations (1):
- Centre for Human and Applied Physiological Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The main data includes videos of participants which are impossible to anonymise. Therefore it is not appropriate for sharing.